CLINICAL TRIAL: NCT02936739
Title: Comparison of Software-assisted Implantation of Elastic Spine Pad (TM) With Respect to Postoperative Change in Neck Disability Index (NDI) With the Conventional Disc Prosthesis Rotaio (TM) After Anterior Cervical Discectomy for Cervical Disc Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCH_ESPvsRotaio
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Intervertebral Disc Displacement
MeSH Terms: conditions — Intervertebral Disc Displacement

ARMS (2):
- Elastic spine pad (Experimental): Patients, who receive Elastic Spine Pad (TM) as cervical disc prosthesis after ventral discectomy.
  Interventions: Device: Anterior cervical discectomy with prosthetic disc replacement / ESP.
- Rotaio (Active Comparator): Patients, who receive Rotaio (TM) as cervical disc prosthesis after ventral discectomy.
  Interventions: Device: Anterior cervical discectomy with prosthetic disc replacement / Rotaio.

INTERVENTIONS:
Device: Anterior cervical discectomy with prosthetic disc replacement / ESP. — Anterior cervical discectomy, with the use of the ESP prosthesis (Manufacturer: FH orthopedics, Mulhouse, France) for the disc replacement.
  Arms: Elastic spine pad
Device: Anterior cervical discectomy with prosthetic disc replacement / Rotaio. — Anterior cervical discectomy, with the use of the Rotaio prosthesis (Manufacturer: Signus Med, Alzenau, Germany) for the disc replacement.
  Arms: Rotaio

SUMMARY:
This is an investigator-initiated study. The primary goal is to evaluate the efficacy of two different cervical disc prosthetic devices with respect to postoperative change in neck disability index. The evaluation will include clinical and radiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Indication for monosegmental anterior cervical discectomy with implantation of a disc prosthesis

Exclusion Criteria:

* Radiologic signs of extensive bone degeneration in the affected segment
* Necessity of implantation of a device smaller in height than 5 mm (as predicted with teh use of the Vertaplan (TM) software
* Transversal spine cord lesion
* Cervical myelopathy
* Preceding surgery on the cervical spine
* Traumatic lesions of the cervical spine
* Radiographic instability in the affected segment: flexion / extension: shift sagittal plane> 3.5 mm or 20% and rotation in the sagittal plane > 20 °, OR in static X-ray examinations: shift in the sagittal plane 3.5 mm or 20% of the vertebral body width and relative sagittal plane angulation > 11º
* signs of instability (Olisthesis) in another segment of the cervical spine
* Active systemic infection
* diseases of the rheumatic type and all autoimmune diseases
* bone metabolic diseases (for example, Paget's disease)
* skeletal metastases
* infections in the cervical spine
* Neurological seizure disorders or other serious neurological disease with risk of falls
* Severe heart failure (NYHA III-IV)
* Bleeding disorders or clopidogrel / coumarins - treatment
* Systemic use of corticosteroids for more than a month in the last 12 months
* Pregnancy
* Legally incompetent patient
* Lactation
* Deformity, anomalies, not fully developed skeleton
* Local tumor disease
* Pre-existing neurologic abnormalities or other shortcomings, such as a Parkinson's disease, diabetic neuropathy, multiple sclerosis, peripheral neuropathy
* Drug / drug or alcohol dependence

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in Neck disability index compared to baseline | 6 weeks, 3, 6, 12 and 24 months postoperative

SECONDARY OUTCOMES:
Change in visual analogue scale for pain in the neck and peripheral pain compared to baseline | 6 weeks, 3, 6, 12 and 24 months postoperative
Change in EuroQOL (EQ-5D) compared to baseline | 6 weeks, 3, 6, 12 and 24 months postoperative
Change in Core Outcome Measure Index (COMI) compared to baseline | 6 weeks, 3, 6, 12 and 24 months postoperative
Change in flexion and extension radiographs compared to baseline | 6 weeks, 3, 6 and 12 months postoperative
Change in and computer aided measurement of segmental height degeneration in adjacent segments compared to baseline | 6 weeks, 3, 6 and 12 months postoperative
Change in consumption of analgetics compared to baseline | 6 weeks, 3, 6, 12 and 24 months postoperative
  The change in analgetics consumption will be assessed on a scale of increase - stable - reduction.
Return to work | 6 weeks postoperative
Return to work | 3 months postoperative
Return to work | 6 months postoperative
Return to work | 12 months postoperative
Return to work | 24 months postoperative
Mortality | 6 weeks postoperative
Mortality | 3 months postoperative
Mortality | 6 months postoperative
Mortality | 12 months postoperative
Mortality | 24 months postoperative
Adverse effects | 6 weeks postoperative
Adverse effects | 3 months postoperative
Adverse effects | 6 months postoperative
Adverse effects | 12 months postoperative
Adverse effects | 24 months postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Uniklinikum Dresden, Dresden, Germany